CLINICAL TRIAL: NCT05508048
Title: The Effects of Existential Approach and Logotherapy Based Psychosocial Support Program on Nursing Students in Period of Pandemic on the Meaning of Life and Life Satisfaction
Brief Title: The Effects of Logotherapy Based Psychosocial Support Program on Nursing Students on the Meaning of Life and Life Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kübra Arslantürk Khalil (Other)
Responsible Party: Sponsor-Investigator, Kübra Arslantürk Khalil, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kübra Arslantürk Khalil
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Meaning of Life and Life Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The existential approach and logotherapy-based psychosocial support program intervention
  Interventions: Behavioral: The existential approach and logotherapy-based psychosocial support program
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: The existential approach and logotherapy-based psychosocial support program — Existential Approach and Logotherapy Based Support Program, which raises awareness about the meaning and purpose of the individual's life, enables them to produce solutions to the sense of meaninglessness, anxiety, feeling of emptiness, and many other problems, and develops different perspectives.The content of the program is base on existential analysis and logotherapy. The program lasted for eight weeks, with the first and last session of the scale applications. Additional sessions were set for each session where the aims and objectives of the session could not achieve. A session lasting at least 50 minutes were held each week.
  Arms: Experimental Group

SUMMARY:
This study is a psychosocial intervention program designed to intervene in the meaning of life and existential problems and life satisfaction in nursing students, especially during the epidemic. In the short term, it expects that students will gain awareness, especially in areas such as life satisfaction, anxiety, aimlessness, the meaning of life, deterioration in functionality, and in the long term, the individual's ultimate issues (death, loneliness, meaning and responsibility) and provide a perspective that can cope with the problems that may arise in these areas. Based on all these, it is aimed to raise awareness of the meaning of life and life satisfaction in nursing students, who constitute a young population, with the existential approach and logotherapy-based psychosocial support program.

H1. The existential approach and logotherapy-based psychosocial support program will affect the experimental group's meaning and purpose of life scale scores.

H2. The existential approach and logotherapy-based psychosocial support program will affect the experimental group's life satisfaction scale scores.

H3. After the existential approach and logotherapy-based psychosocial support program, there will be a significant difference between the experimental and control groups' meaning and purpose of life scores.

H4. After the existential approach and logotherapy-based psychosocial support program, there will be a significant difference between the experimental and control groups' life satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Completed mental health and psychiatric nursing course
* Agreeing to participate as a result of the research announcement
* No acute psychiatric problem
* Those who have not lost their first-degree relative due to Covid-19

Exclusion Criteria:

* Having an acute psychiatric problem
* Those who lost their first-degree relative due to Covid-19

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Group Difference-Meaning and Purpose | 10 weeks
  A statistically significant difference was determined in terms of the last measurement MPLS-total scores according to the groups.
Between Groups Difference-Life Satisfaction | 10 weeks
  A statistically significant difference was found in terms of the last measurement life satisfaction scale scores according to the groups.
In Group Difference-Life Satisfaction | 10 weeks
  A statistically significant difference was found in the first measurement - last measurement life satisfaction scale scores of the experimental group.
In Group Difference-Meaning and Purpose | 10 weeks
  A statistically significant difference was found in the first measurement - last measurement MPLS- total scores of the experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No